CLINICAL TRIAL: NCT01579201
Title: ED90 Determination of Carbetocin for the Prevention of Postpartum Uterine Atony in Women Undergoing an Elective Cesarean Delivery
Brief Title: ED90 Determination of Carbetocin for the Prevention of Uterine Atony in Women Undergoing an Elective Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Christian Loubert, Christian Loubert, MD, FRCPC, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: LoubertHMR2012/01
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Postpartum Hemorrhage; Uterine Atony
Keywords: Postpartum Hemorrhage; Uterine Atony; Obstetric Anesthesia; Cesarean Section; Carbetocin
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia | interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carbetocin (Experimental)
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — First patient: 70 mcg. Following doses according to biased coin design up-down sequential allocation method, with increments or decrements of 10 mcg. An unsatisfactory uterine tone will lead to an increment while a satisfactory uterine tone will result in either a decrement or no change.
  Other Names: Duratocin

SUMMARY:
The purpose of this trial is to determine the effective dose of carbetocin which would prevent the occurrence of postpartum uterine atony in 90% of women undergoing an elective cesarean delivery.

DETAILED DESCRIPTION:
Postpartum hemorrhage is a major cause of maternal morbidity and mortality worldwide. Carbetocin have been shown effective in the prevention of uterine atony, which is the leading cause of postpartum hemorrhage. The Society of Obstetricians and Gynecologists of Canada recommends a single 100 mcg dose of carbetocin after elective cesarean delivery to prevent postpartum hemorrhage. However, there is no clear data in the literature regarding the lowest effective dose of carbetocin that should be administered. The use of the minimum effective dose of carbetocin may reduce its side effects, including hypotension, tachycardia, nausea, vomiting and flushing.

In this trial, healthy term pregnant women undergoing elective cesarean delivery under spinal anesthesia will be recruited. The effective dose of carbetocin that will prevent postpartum uterine atony in 90% of the women (ED90) will be determined using a biased coin design up-down sequential allocation method. The determination of the carbetocin ED90 will help the anesthesiologist regarding the optimal dose of carbetocin to administer after elective cesarean delivery to prevent uterine atony.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women (ASA I or II)
* Elective cesarean delivery
* Spinal anesthesia
* Term gestation (37 weeks and above)

Exclusion Criteria:

* Multiple gestation
* Known coagulopathy
* Active labour
* Uterine fibroids
* Body mass index > 45
* Emergency cesarean section
* General anesthesia
* Any contraindication to neuraxial anesthesia
* Cardiopathies
* Known allergies to carbetocin
* Patient refusal
* Placenta previa/Placenta accreta
* Hypertensive disease/Preeclampsia/Eclampsia
* Polyhydramnios
* Previous history of uterine atony or postpartum hemorrhage
* Renal or liver disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Dose of carbetocin which will prevent uterine atony in 90% of subjects | 5 minutes
  The uterine tone will be assessed by the obstetrician by palpation 5 minutes after injection. The uterine tone will be judged either as satisfactory or unsatisfactory.

SECONDARY OUTCOMES:
Incidence of side effects | 20 minutes
  Any of these side effects will be noted in the first 20 minutes following injection of carbetocin: hypotension, tachycardia, nausea, vomiting, flushing, headache, feeling of warmth, tremor, metallic taste, abdominal pain, back pain, chest pain and others.
Vasopressors administered | 20 minutes
  The total dose of vasopressors administered in the first 20 minutes following the administration of carbetocin will be noted.
Anti nausea therapy | 20 minutes
Additional uterotonic medication administered | 20 minutes
Additional uterine massage | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Christian Loubert, MD, FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada